CLINICAL TRIAL: NCT00790881
Title: Pharmacokinetic Interaction Between the Antimalarial Combination Artemether/Lumefantrine and Combination Antiretroviral Therapy Including Nevirapine in HIV-infected Adults
Brief Title: Artemether/Lumefantrine and Nevirapine Interaction Study in HIV-infected Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Cape Town (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other)
Responsible Party: ACT Consortium, London School of Hygiene & Tropical Medicine
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SEACAT 2.4.1; DOH-27-0807-2012
Record Dates: First submitted 2008-11-13; First posted 2008-11-14 (Estimated); Last update posted 2010-06-28 (Estimated); Status verified 2010-06

CONDITIONS: Malaria; HIV
Keywords: malaria; HIV; AIDS; nevirapine; lumefantrine; artemether; drug interaction; pharmacokinetics
MeSH Terms: conditions — Malaria; Acquired Immunodeficiency Syndrome | interventions — Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Antiretroviral-naive (Other): Antiretroviral-naive included as control group
  Interventions: Drug: Artemether/Lumefantrine
- Nevirapine-based antiretroviral therapy (Active Comparator): Nevirapine-based antiretroviral therapy
  Interventions: Drug: Artemether/ lumefantrine

INTERVENTIONS:
Drug: Artemether/Lumefantrine — Coartem (fixed dose Artemether20mg /Lumefantrine 120mg) Dose: 4 tablets(80mg/480mg) twice daily for 3 days at 0,8,24,36,48 and 60 hours
  Other Names: Coartem
  Arms: Antiretroviral-naive
Drug: Artemether/ lumefantrine — Coartem (fixed dose Artemether20mg /Lumefantrine 120mg) Dose: 4 tablets(80mg/480mg) twice daily for 3 days at 0,8,24,36,48 and 60 hours
  Other Names: Coartem
  Arms: Nevirapine-based antiretroviral therapy

SUMMARY:
Despite the clinical significance of potential interactions between antimalarials and antiretrovirals, no drug interaction studies have been published and there is an urgent need to address this gap in current knowledge.

This study aims to assess the drug interaction between the antimalarial Artemether/Lumefantrine used for management of uncomplicated malaria and Nevirapine-based antiretroviral therapy.

ELIGIBILITY:
Inclusion Criteria:

* Informed and given ample time and opportunity to think about participation and willing and able to comprehend and comply with all trial requirements. The participant has given written informed consent to participate in the study and to abide by study restrictions.
* Male or female subjects older than 18 years of age.
* HIV-infected as documented by positive HIV-antibody test and confirmed by Western blot.
* Body weight more than 35kg with a body mass index (BMI) ranging between 18.5 to 30kg/m2 inclusive (See Appendix 16.2).
* Karnofsky score above 70 (See Appendix 16.5).
* CD4 count ≥ 200 cells/mm3
* Patients on NVP-based cART at stable doses without significant toxicity for at least 6 weeks at screening (Group 2 only).

Exclusion Criteria:

* Patients diagnosed with Plasmodium falciparum malaria
* Contraindications to artemether/lumefantrine:

  * Hypersensitivity to the artemether, lumefantrine or to any of the excipients of Coartem®.
  * Patients with severe malaria according to WHO definition.
  * Pregnant (as confirmed by an HCG test performed at screening) or breast-feeding female.
  * Patients with a family history of congenital prolongation of the QTc interval or sudden death or with any other clinical condition known to prolong the QTc interval such as patients with a history of symptomatic cardiac arrhythmias, with clinically relevant bradycardia or with severe cardiac disease.
  * Patients with known disturbances of electrolyte balance e.g. hypokalaemia or hypomagnesaemia.
  * Patients taking any drug which is metabolised by the cytochrome enzyme CYP2D6 (e.g. flecainide, metoprolol, imipramine, amitriptyline, clomipramine).
  * Patients taking drugs that are known to prolong the QTc interval such as antiarrhythmics of classes IA and III, neuroleptics, antidepressive agents, certain antibiotics including some agents of the following classes: macrolides, fluoroquinolones, imidazole, and triazole antifungal agents, certain non-sedating antihistaminics (terfenadine, astemizole), cisapride.
* Contraindication to nevirapine:

  * Hypersensitivity to nevirapine or any of the excipients of Aspen Nevirapine®.
  * Severe hepatic dysfunction: Child-Pugh class B or C and in endstage renal failure in patients not on haemodialysis.
  * Aspartate transaminase (AST) or alanine aminotransferase (ALT) > 5 x upper limit of normal (ULN).
  * History of severe rash, rash accompanied by constitutional symptoms; hypersensitivity syndrome, or clinical hepatitis due to nevirapine.
* Haemoglobin below 8.5g/dL for female and 9.5g/dL for male subjects.
* Pharmacokinetic exclusion criteria:

  * Relevant history or current condition(s) that might interfere with drug absorption, distribution, metabolism or excretion.
  * Current smokers, or subjects who have stopped smoking less than 3 months prior to the date of screening.
  * History of or current substance abuse problem or a positive urine screen for drugs of abuse.
  * History of or current compulsive alcohol abuse problem.
  * The subject has consumed any alcohol, grapefruit or caffeine-containing products (ie tea, coffee, cola, chocolate) within 24 hours before the first dose of AL during each PK profile.
  * The subject has participated in strenuous exercise within 24 hours before the first IP administration.
* General exclusion criteria:

  * Severely ill or suffering from any serious underlying disease (particularly cardiac, hepatic or renal disease) that in the opinion of the Investigator would make the participant unsuitable for the study in terms of their safety or study analysis.
  * The volunteer has participated in another study with any investigational product within 8 weeks before the first administration of the current investigational products, or until at least 5 x t½ elimination has lapsed, whichever is the greater.
  * Subjects who, in the opinion of the Investigator, should not participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-08 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Lumefantrine plasma concentration | day 7

SECONDARY OUTCOMES:
Point estimates and 90% confidence intervals for the mean ratios of the lumefantrine, artemether and DHA log-transformed Cmax, AUC0-t, AUC0 ∞ , t½,z, tmax and MRT with/without NVP | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Karen Barnes, MD, Principal Investigator — University of Cape Town; Tamara Kredo, MD, Study Director — University of Cape Town
Locations (1):
- Groote Schuur Hospital, Research ward, Cape Town, South Africa

REFERENCES:
- [Derived] Kredo T, Mauff K, Van der Walt JS, Wiesner L, Maartens G, Cohen K, Smith P, Barnes KI. Interaction between artemether-lumefantrine and nevirapine-based antiretroviral therapy in HIV-1-infected patients. Antimicrob Agents Chemother. 2011 Dec;55(12):5616-23. doi: 10.1128/AAC.05265-11. Epub 2011 Sep 26. PMID 21947399